CLINICAL TRIAL: NCT06510959
Title: ACTIVE Ageing in Changing Societies. Older People's Social and Digital Resources in Pandemic and Post-pandemic ITaly (ACTIVE-IT). Research Stream 3 - Older People, New Needs, and Possible Solutions. A Pilot Study on Peer-to-peer Digital Education
Brief Title: Older People, New Needs, and Possible Solutions. A Pilot Study on Peer-to-peer Digital Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: University of Pavia (Other); University of Applied Sciences and Arts of Southern Switzerland (Other); Catholic University, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-0897
Record Dates: First submitted 2024-06-05; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Well-Being, Psychological; Digital Skills
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital course (Other): 10-lesson weekly course taught by a peer on the use of smartphones and daily utility apps.
  Interventions: Other: Digital course

INTERVENTIONS:
Other: Digital course — The course aims to enhance participants' digital skills concerning the use of smartphones, specifically focusing on daily utility apps such as email apps, eGov apps, mobility apps, etc. The course is structured into the following ten 90-minute weekly lessons.

SUMMARY:
"Older people, new needs, and possible solutions: A pilot study on peer-to-peer digital education" aims to create a digital literacy protocol targeted specifically to older people, providing them with the digital skills needed to age healthily and actively in a changing social context. Specifically, the main goal is to pilot (by designing, implementing, and evaluating) a peer-to-peer digital literacy course, whereby older educators teach less digitally savvy older people how to use smartphone daily utility apps, such as e-Gov, home banking, etc.

To evaluate the effect of the intervention on participants, smartphone usage patterns are measured before, during, and after the course. Then, the impact of the course on participants' perception of well-being is assessed as well.

DETAILED DESCRIPTION:
This study aims to pilot, by designing, implementing, and evaluating, a digital peer education course for older people, focusing specifically on the use of smartphones and daily utility apps. The course has been co-designed with AUSER MB, a non-profit organization involved in active aging, and the peer tutors. It is structured in ten 90-minute classes covering topics such as emails, online accounts, app downloads, e-Gov apps, healthcare apps, mobility and payment apps, etc. The 30 participants, divided into three groups, have been selected among the 65+ year-old people attending the computer classes already offered by AUSER MB and having a personal smartphone, as a very basic set of digital skills and familiarity with digital devices was necessary for the slightly more advanced topics covered by the course.

In addition to piloting the course and aiming to define a protocol that could be replicated in other similar contexts, this study aims to measure the effect of the course on participants' digital skills and their perceived well-being. To do so, the investigators adopted a mixed methods approach, employing digital methods by collecting and analyzing data on participants' smartphone use (i.e., log data on smartphone use before/during/after the intervention), a quasi-experiment collecting information on course participants' well-being before/after the course attendance using a questionnaire survey, and ethnographic observation conducted during the course, observing interactions between subjects during the course.

The study is part of the project "ACTIVE ageing in changing societies. Older people's social and digital resources in pandemic and post-pandemic Italy (ACTIVE-IT)", funded by the Italian Fondazione Cariplo

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older
* personal smartphone

Exclusion Criteria:

* N/A

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Smartphone usage patterns | Four months (feb 24 - jun 24)
  To evaluate changes in smartphone usage patterns, the investigators collect smartphone usage data for about four months: (one month) before the start of the course, during the course attendance, and (one month) after the course has ended through the app Stay Free - Screen Time. This app collects the categories of the apps that participants used during the monitoring period, the exact time (day, hour, minutes) the apps started/stopped to be used, and the duration (in seconds) of use of each apps' category. The category of the apps and the duration of use, as well as the day in which they have been used, will be combined to study participants' using habits.
Perception of wellbeing | Two measurements: baseline, pre-intervention and immediately after the intervention
  To evaluate the impact of the peer-to-peer digital education course on participants' wellbeing, the investigators will adopt a quasi-experiment approach, inviting course participants to fill in a short online self-completed questionnaire during the first and last class of the course. The investigators will collect the following five types of measures: current use of and competence on digital device use, attitudes towards technology, life satisfaction, happiness and wellbeing, demographic and socio-economic characteristics, health status.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milan - Bicocca, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymised qualitative and quantitative data will be deposited within the UniData Bicocca Data Archive.
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: Website of the research group — https://ageingsocieties.unimib.it/